CLINICAL TRIAL: NCT03358836
Title: Joint Health Study
Status: Completed | Type: Observational
Sponsor: Bloodworks (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: Joint Health Study
Record Dates: First submitted 2017-11-25; First posted 2017-12-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; FIX; Factor IX; Factor 9
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will draw up to 40 mL (3 tablespoons) of blood to test for factor level, inhibitor level, and biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Episodic treatment with FIX concentrates for bleeding episodes
- Group B: Prophylaxis using any FIX concentrate with an intended trough of 1-5%
- Group C: Prophylaxis with an extended half-life (EHL) FIX with an intended trough of >10%

SUMMARY:
This is a prospective, non-randomized, controlled study to examine whether or not having a higher trough during prophylactic treatment with clotting factor offers better joint protection than the standard trough of 1% Factor IX (FIX or Factor 9). This study will test the hypothesis that an extended half-life (EHL) FIX product with an intended trough of >10% could offer better protection than previous treatment concentrates. This study also examines whether or not joint damage could be diagnosed earlier using ultrasound images.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, controlled study to examine whether or not having a higher trough during prophylactic treatment with clotting factor offers better joint protection than the standard trough of 1% Factor IX (FIX or Factor 9). This study will test the hypothesis that an extended half-life (EHL) FIX product with an intended trough of >10% could offer better protection than previous treatment concentrates. This study also examines whether or not joint damage could be diagnosed earlier using ultrasound images. The primary research question is whether EHL rIX with an intended trough level of >10% will improve the outcome of joint health of elbow, ankle, and knee joints as assessed with ultrasound assessments in patients with severe Hemophilia B.

Depending on their current treatment regimen, subjects will be in one of three groups: 1) on demand, 2) prophylaxis with an intended trough of 1-5%, and 3) prophylaxis with an intended trough of >10%. Subjects will have four annual study visits over three years: baseline, year 1, year 2, and year 3. At each of these visits, subjects will complete questionnaires, joint assessments, have their blood taken, and have ultrasound images of their joints. The first 10 subjects will also have x-rays and MRIs of their joints for ultrasound validation.

Subjects are encouraged to come in during a painful episode for an examination, assessment, and ultrasound of their joints and to come in again within 1-2 weeks after the painful episode for a repeat examination, assessments, and ultrasound.

This study will be conducted at the Washington Center for Bleeding Disorders (WCBD) at Bloodworks Northwest, Oregon Health & Science University (OHSU), University of California San Diego (UCSD), University of California Los Angeles (UCLA), and Tulane University (TU). Cumulatively across the five sites, up to 50 participants will be enrolled. Additional sites may be added.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia B (FIX <1%)
* Either on demand or on prophylaxis with rFIX or EHL-rIX products with the intention to stay on the current regimen for the next 3 years
* For Group C, start of this treatment regimen up to 6 months prior is permissible

Exclusion Criteria:

* Other known bleeding disorder
* Other rheumatologic disorder affecting joints
* Other known neuromotor defect (making physical exam difficult)

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants are male, age 16 or older, have severe hemophilia B, and are currently on either an episodic or prophylactic treatment regimen with FIX concentrates
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Joint health status | Change from baseline at up to three years
  Joint health status in all six major joints (elbows, knees, and ankles) in all three groups as assessed by ultrasound

SECONDARY OUTCOMES:
Joint and overall health status | Change from baseline at up to three years
  Observational assessment of joint and overall health status evaluated by activity level, functional assessment, pain assessment, joint examination, and adherence
Joint health at year 1 | Change from baseline at up to one year
  Observational assessment of joint health at year one in the different groups
Joint health at year 2 | Change from baseline at up to two years
  Observational assessment of joint health at year two in the different groups
Acute events/bleeding | Change from baseline at up to three years
  Observational assessment of ultrasound findings during acute events/bleeding with an opportunity to follow longitudinally to gain understanding of natural evolution of bleeding as shown by ultrasound
Biomarkers | Change from baseline at up to three years
  Exploration of potential biomarkers for joint health

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kruse-Jarres, MD, MPH, Principal Investigator — Washington Center for Bleeding Disorders at Bloodworks Northwest
Locations (5):
- United States (5):
  - Orthopaedic Institute for Children at University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Tulane University, New Orleans, Louisiana
  - Oregon Health & Science University, Portland, Oregon
  - Washington Center for Bleeding Disorders at Bloodworks Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03358836/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Form (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03358836/ICF_001.pdf
  • Informed Consent Form: Assent Ages 16 to 17 (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03358836/ICF_002.pdf